CLINICAL TRIAL: NCT02375555
Title: An Open-Label, Single Arm, Phase 2a Study of Bortezomib, Lenalidomide, Dexamethasone and Elotuzumab in Newly Diagnosed Multiple Myeloma
Brief Title: Study of Bortezomib,Lenalidomide,Dexamethasone & Elotuzumab in Newly Diagnosed MM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Jacob Laubach, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-453
Record Dates: First submitted 2015-01-13; First posted 2015-03-02 (Estimated); Results first posted 2023-12-06 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; elotuzumab; Bortezomib; Dexamethasone; Calcium Dobesilate; Hematopoietic Stem Cell Mobilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Elotuzumab, lenalidomide, bortezomib, and dexamethasone (Experimental): Participants will receive therapy with the combination of lenalidomide, bortezomib, and dexamethasone and elotuzumab (E-RVD). Induction cycles (1 to 8) are 21-day cycles.
  * Elotuzumab will be administered by intravenous (IV) infusion
  * Bortezomib as a subcutaneous injection
  * Lenalidomide single daily oral dose
  * Dexamethasone as oral tablets and IV infusion
  * Stem cell mobilization will be performed for all subjects at the end of Cycle 4.
  Subjects may elect to stop E-RVD at the end of Induction Cycle 4 and proceed to autologous SCT. Subjects who do not proceed to SCT may receive a full 8 cycles of induction therapy.
  The maintenance schedule (28 days) will start after 8 cycles of induction regimen for subjects not proceeding with SCT, or after recovery from SCT for subjects proceeding with it.
  Maintenance therapy with E-RVD will be administered to all patients, with the specific maintenance regimen determined by risk category.
  Interventions: Drug: Lenalidomide; Drug: Elotuzumab; Drug: Bortezomib; Drug: Dexamethasone; Procedure: Stem Cell Mobilization

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: Revlimid®
Drug: Elotuzumab
  Other Names: HuLuc63
Drug: Bortezomib
  Other Names: Velcade
Drug: Dexamethasone
  Other Names: Baycadron Elixer; Decadron
Procedure: Stem Cell Mobilization

SUMMARY:
This research study is evaluating a combination of four drugs -- lenalidomide, bortezomib, dexamethasone and elotuzumab -- as therapy for newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial testing the safety and effectiveness of an investigational drug (in this case elotuzumab) in combination with lenalidomide, bortezomib and dexamethasone to learn more about the side effects of this regimen and whether it is effective in newly diagnosed multiple myeloma.

"Investigational" means that the drug elotuzumab and the combination of this agent with lenalidomide, bortezomib, and dexamethasone are being studied. It also means that the the U.S. Food and Drug Administration (FDA) has not yet approved elotuzumab for the treatment of cancer. The drugs, lenalidomide, bortezomib, and dexamethasone are approved by the FDA. Participants in this trial will have the option to undergo autologous stem cell transplantation (ASCT) following initial therapy with elotuzumab, lenalidomide, bortezomib, and dexamethasone. ASCT is a standard of care in the treatment of multiple myeloma. All participants, including those who undergo ASCT and those who choose not to, will receive what is referred to as "maintenance therapy" - or continuous treatment - after the initial cycles of treatment with elotuzumab, lenalidomide, bortezomib, and dexamethasone. The specific maintenance regimen will be determined by risk category.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria on screening examination to be eligible to participate in the study. All laboratory assessments should be performed within 21 days of initiation of protocol therapy unless otherwise specified.Subject is, in the investigator's opinion, willing and able to comply with the protocol requirements.
* Subject has given voluntary signed written informed consent before performance of any study-related procedure that is not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to their future medical care.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (see Appendix 1).
* Subject is a candidate for high-dose therapy and autologous SCT based on standard criteria at the institution where this treatment will be administered.
* Newly diagnosed untreated, symptomatic, documented MM based on standard diagnostic criteria (Rajkumar 2009) with measurable disease, defined as any of the following:

  * Serum Immunoglobulin G (IgG), Immunoglobulin (A) IgA, or Immunoglobulin M (IgM) M-protein ≥ 0.5 g/dL, or
  * Serum Immunoglobulin D (IgD) M-protein ≥ 0.05 g/dL, or
  * Urinary M-protein excretion of more than 200 mg/24 hours, or
  * Serum free light chains (FLC) of at least 100 mg/dL with an abnormal FLC ratio
* Subject agrees to refrain from blood donations during therapy on study and for 8 weeks after therapy is completed.
* Men and women, age ≥18 years or legal age of consent per local regulations (whichever is greater).
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting Lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking Lenalidomide through 90 days after the last dose of study drug. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy from the time of signing the informed consent form through 90 days after the last dose of study drug. All patients must be registered in and must comply with all requirements of the Revlimid Rems™ program.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Diagnosed with smoldering MM, monoclonal gammopathy of undetermined significance, Waldenstrom's macroglobulinemia, Plasma cell leukemia, POEMS syndrome or amyloidosis.
* Participant has ≥ Grade 2 peripheral neuropathy on clinical examination within 21 days before initiation of protocol therapy.
* Renal insufficiency, defined as creatinine clearance < 30 mL/min (either actual or calculated value), within 21 days of initiation of protocol therapy. The Cockgroft-Gault formula should be used for calculating creatinine clearance values:

  * (140-age) x Body mass (kg) x 0.85 (female) or 1.0 (male) serum creat (mg/dL) x 72
  * Ideal body weight (IBW) should be used if actual body weight is > 20% above IBW
* Platelet count <75,000 cells/mm3 at time of screening evaluation. Transfusion may not be used to meet platelet eligibility criteria within 7 days of obtaining screening evaluation.
* Participants with an absolute neutrophil count (ANC) < 1000 cells/mm3 at time of screening evaluation. Growth factor may not be used to meet ANC eligibility criteria within 14 days of obtaining screening evaluation.
* Participants with hemoglobin level < 8.0 g/dL, at time of screening. Transfusion may not be used to meet eligibility criteria within 7 days of obtaining screening evaluation.
* Participants with hepatic impairment, defined as bilirubin > 1.5 x institutional upper limit of normal (ULN) or AST (Aspartate aminotransferase; SGOT), ALT (Alanine aminotransferase; SGPT), or alkaline phosphatase > 3x institutional ULN, within 21 days of initiation of protocol therapy
* Other ongoing or prior anti-myeloma therapy. Patients may be receiving concomitant therapy with bisphosphonates and low dose corticosteroids (e.g., prednisone up to but no more than 10 mg p.o. q.d. or its equivalent) for symptom management and comorbid conditions. Doses of corticosteroid should be stable for at least 7 days prior to study treatment.)
* Known significant cardiac abnormalities including:

  * Congestive heart failure, New York Heart Association (NYHA) class III or IV
  * Uncontrolled angina, arrhythmia or hypertension
  * Myocardial infarction within the past six months
  * Any other uncontrolled or severe cardiovascular condition
  * Prior cerebrovascular event with residual neurologic deficit
* Serious, intercurrent illness including, but not limited to, clinically relevant active infection, known active hepatitis B or C viral infection, known HIV infection, uncontrolled diabetes mellitus, or serious co-morbid medical conditions such as chronic restrictive pulmonary disease, and cirrhosis.
* Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at unacceptable risk if he/she were to participate in the study.
* Prior malignancy (within the last 5 years) except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* Known hypersensitivity to acyclovir or similar anti-viral drug
* Known intolerance to steroid therapy
* Contraindication or prior intolerance to thromboembolic prophylaxis with aspirin, warfarin or low-molecular weight heparin
* Participants with known brain metastases.
* Poor tolerability or known allergy to any of the study drugs or compounds of similar chemical or biologic composition to dexamethasone, boron or mannitol.
* Female participants pregnant or breast-feeding.
* Participants who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of the surgery.
* Participants with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob P. Laubach, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Levine Cancer Institute, Charlotte, North Carolina
  - Virginia Cancer Specialists, Fairfax, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from May 2015 to April 2016.
Groups:
- Elotuzumab, Lenalidomide, Bortezomib, and Dexamethasone: Participants will receive therapy with the combination of lenalidomide, bortezomib, and dexamethasone and elotuzumab (E-RVD). Induction cycles (1 to 8) are 21-day cycles.
  * Elotuzumab will be administered by intravenous (IV) infusion
  * Bortezomib as a subcutaneous injection
  * Lenalidomide single daily oral dose
  * Dexamethasone as oral tablets and IV infusion
  * Stem cell mobilization will be performed for all subjects at the end of Cycle 4.
  Subjects who attain at least a partial response (PR) may elect to stop E-RVD at the end of Induction Cycle 4 and proceed to autologous SCT. Subjects who do not proceed to SCT may receive 8 cycles of induction therapy.
  - The maintenance schedule (28 days) will start after 8 cycles of induction regimen for subjects not proceeding with SCT, or after recovery from SCT for subjects proceeding with it.
  Maintenance therapy with E-RVD will be administered to all patients, with the specific maintenance regimen determined by risk category.
  Lenalidomide
  Elotuzumab
  Bortezomib
  Dexamethasone
  Stem Cell Mobilization
Period: Induction Period
Arm/Group | Elotuzumab, Lenalidomide, Bortezomib, and Dexamethasone
Started | 40
Induction Therapy Cycles 1-4 | 34 (Of the 40 patients comprising the safety population, 34 patients completed 4 cycles (cycles 1-4) of induction therapy.)
Induction Therapy Cycles 5-8 | 12 (Of the 40 patients comprising the safety population, 12 patients completed 4 additional cycles (cycles 5-8) of induction therapy.)
Autologous Stem Cell Transplant | 19 (Of the 40 patients comprising the safety population, 19 patients received autologous stem cell transplant (ASCT) at the end of Induction cycle 4.)
Completed | 29
Not Completed | 11
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 2
Not completed — Other | 1
Not completed — Didn't meet criteria for maintenance therapy | 1
Period: Maintenance Period
Arm/Group | Elotuzumab, Lenalidomide, Bortezomib, and Dexamethasone
Started | 29
Completed | 0
Not Completed | 29
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 4
Not completed — Death | 1
Not completed — Disease Progression | 5
Not completed — Patient Non-compliance | 1
Not completed — Still on maintenance | 16

BASELINE CHARACTERISTICS:
Population: The analysis population is safety- all treated participants.
Groups:
- Elotuzumab, Lenalidomide, Bortezomib, and Dexamethasone: Participants will receive therapy with the combination of lenalidomide, bortezomib, and dexamethasone and elotuzumab (E-RVD). Induction cycles (1 to 8) are 21-day cycles.
  * Elotuzumab will be administered by intravenous (IV) infusion
  * Bortezomib as a subcutaneous injection
  * Lenalidomide single daily oral dose
  * Dexamethasone as oral tablets and IV infusion
  * Stem cell mobilization will be performed for all subjects at the end of Cycle 4.
  Subjects may elect to stop E-RVD at the end of Cycle 4 and proceed to autologous SCT. Subjects who do not proceed to SCT may receive 8 cycles of induction therapy.
  The maintenance schedule (28 days) will start after 8 cycles of induction regimen for subjects not proceeding with SCT, or after recovery from SCT for subjects proceeding with it.
  Maintenance therapy with E-RVD will be administered to all patients, with the specific maintenance regimen determined by risk category.
Arm/Group | Elotuzumab, Lenalidomide, Bortezomib, and Dexamethasone
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 6
  White | 28
  More than one race | 0
  Unknown or Not Reported | 5
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status: (PS0) Fully active, able to carry on all pre-disease performance without restriction (PS1) Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (PS2) Ambulatory and capable of all self-care but unable to carry out any work activities; Up and about >50% of waking hours. Higher grades indicate more severe disease.
  Participants
    Grade 0 | 26
    Grade 1 | 13
    Grade 2 | 1
International Staging System (ISS) Multiple Myeloma Stage [Count of Participants; unit: Participants] — The International Staging System (ISS) consists of three stages: stage I, serum beta 2-microglobulin level lower than 3.5 mg per liter and serum albumin level 3.5 g per deciliter or higher; stage II, neither stage I nor III; and stage III, serum beta 2-microglobulin level 5.5 mg per liter or higher. Higher stages indicate more severe disease.
  Participants
    Stage I | 24
    Stage II | 10
    Stage III | 6
Cytogenetic risk classification [Count of Participants; unit: Participants] — Bone marrow aspiration and biopsy to be evaluated for cytogenetics by standard banding and FISH, including marrow karyotyping if possible. High-risk cytogenetics include presence of translocations t(4;14), t(14;16) or del17p.
  Participants
    High | 6
    Standard | 19
    Missing | 15

OUTCOME MEASURES:

1. Primary Outcome: 4 Cycle Response Rate
Description: Disease response was defined as the proportion of patients who achieved a response of partial response or better using International Myeloma Working Group (IMWG) response criteria. Partial Response (PR) defined as 50% reduction of serum M-protein and reduction in 24h urinary M-protein by ≥90% or to <200mg/24h; Very Good Partial Response (VGPR) defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein plus urine M-protein level <100mg/24h; Complete Response (CR) defined as negative immunofixation on serum and urine and, disappearance of any soft tissue plasmacytomas and, <5% plasma cells in BM; Stringent Complete Response (sCR) defined as normal FLC ratio and absence of clonal cells in BM by immunohistochemistry or 2-4 color flow cytometry. The Clopper and Pearson method was used to estimate the 95% CIs for the response rate at Week 12.
Time Frame: Participants were followed up to 12 weeks.
Population: The analysis dataset is comprised of 34 efficacy-evaluable participants, where it was defined as participants who were dosed, had a post-baseline scan and also had at least 4-cycles of induction.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Elotuzumab, Lenalidomide, Bortezomib, and Dexamethasone
Number analyzed (Participants) | 34
proportion of participants | 0.971 [0.847 to 0.999]

2. Secondary Outcome: Successful Stem Cell Mobilization (SC Mob) Rate
Description: Successful SC Mob defined as the proportion of participants with the ability to collect a total of at least 2*10^6 CD34+ cells/kg.
Time Frame: The most distant time of stem cell mobilization from time of registration is 21.4 weeks with a median of 15.14 weeks.
Population: The analysis population is comprised of participants who underwent stem cell mobilization after completing 4 cycles of induction therapy.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Elotuzumab, Lenalidomide, Bortezomib, and Dexamethasone
Number analyzed (Participants) | 31
proportion of participants | 0.968 [0.833 to 0.999]

3. Secondary Outcome: 4 Cycle Ever Dose Modification (DM) Rate
Description: The 4 cycle ever DM rate is the proportion of participants who started therapy and required dose modification of any study drug during the first four cycles of E-RVD.
Time Frame: Participants were followed up to 12 weeks.
Population: The analysis dataset is comprised of participants who were dosed (parallel with the safety population).
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Elotuzumab, Lenalidomide, Bortezomib, and Dexamethasone
Number analyzed (Participants) | 40
proportion of participants | .40 [.25 to .57]

4. Secondary Outcome: Grade 3 and 4 Treatment-Emergent Adverse Event (TEAE) Rate
Description: Grade 3 and 4 TEA rate was defined as the proportion of participants who experienced a grade 3 or 4 adverse event of any attribution based on NCI Common Toxicity Criteria for Adverse Events Version 4 (CTCAEv4) on treatment.
Time Frame: The adverse event observation period defined as the time on treatment (+30d) is 278 weeks.
Population: All participants in the safety population.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Elotuzumab, Lenalidomide, Bortezomib, and Dexamethasone
Number analyzed (Participants) | 40
proportion of participants | 0.70 [0.53 to 0.83]

5. Secondary Outcome: Best Responses to E-RVD.
Description: Best responses to E-RVD was assessed using International Myeloma Working Group (IMWG) response criteria: Partial Response (PR) defined as 50% reduction of serum M-protein and reduction in 24h urinary M-protein by ≥90% or to <200mg/24h; Very Good Partial Response (VGPR) defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein plus urine M-protein level <100mg/24h; Complete Response (CR) defined as negative immunofixation on serum and urine and, disappearance of any soft tissue plasmacytomas and, <5% plasma cells in BM; Stringent Complete Response (sCR) defined as normal FLC ratio and absence of clonal cells in BM by immunohistochemistry or 2-4 color flow cytometry.
Time Frame: Participants were followed up to 273.6 weeks.
Population: Best responses to E-RVD in the safety population, defined as participants with Multiple Myeloma who received one or more dose of elotuzumab. Out of the 40 participants included in the safety population, one participant did not receive or more dose of elotuzumab, and was not included in the best response analysis population.
Measure: Count of Participants; unit: Participants
Groups:
- All Patients Treated With E-RVD (40 Patients).: Participants will receive therapy with the combination of lenalidomide, bortezomib, and dexamethasone and elotuzumab (E-RVD). Induction cycles (1 to 8) are 21-day cycles.
  * Elotuzumab will be administered by intravenous (IV) infusion
  * Bortezomib as a subcutaneous injection
  * Lenalidomide single daily oral dose
  * Dexamethasone as oral tablets and IV infusion
  * Stem cell mobilization will be performed for all subjects at the end of Cycle 4.
  Subjects may elect to stop E-RVD at the end of Cycle 4 and proceed to autologous SCT. Subjects who do not proceed to SCT may receive 8 cycles of induction therapy.
  The maintenance schedule (28 days) will start after 8 cycles of induction regimen for subjects not proceeding with SCT, or after recovery from SCT for subjects proceeding with it.
  Maintenance therapy with E-RVD will be administered to all patients, with the specific maintenance regimen determined by risk category.
Arm/Group | All Patients Treated With E-RVD (40 Patients).
Number analyzed (Participants) | 39
Participants
  Sustained complete response (sCR) | 9
  Complete response (CR) | 8
  Very good partial response (VGPR) | 16
  Partial response (PR) | 5
  Minimal response (MR) | 1

6. Secondary Outcome: Objective Response Rate (ORR) at End of 8 Cycles of Induction Therapy.
Description: ORR was defined as the proportion of patients who achieved a disease response of partial response (PR) or better using IMWG response criteria. PR defined as 50% reduction of serum M-protein and reduction in 24h urinary M-protein by ≥90% or to <200mg/24h; Very Good Partial Response (VGPR) defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein plus urine M-protein level <100mg/24h; Complete Response (CR) defined as negative immunofixation on serum and urine and, disappearance of any soft tissue plasmacytomas and, <5% plasma cells in BM; Stringent Complete Response (sCR) defined as normal FLC ratio and absence of clonal cells in BM by immunohistochemistry or 2-4 color flow cytometry.
Time Frame: Participants were followed up to 24 weeks.
Population: Safety population comprised of 40 patients, of which 19 received ASCT and 12 completed 8 full induction cycles.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- All Patients Treated With E-RVD.: Participants will receive therapy with the combination of lenalidomide, bortezomib, and dexamethasone and elotuzumab (E-RVD). Induction cycles (1 to 8) are 21-day cycles.
  * Elotuzumab will be administered by intravenous (IV) infusion
  * Bortezomib as a subcutaneous injection
  * Lenalidomide single daily oral dose
  * Dexamethasone as oral tablets and IV infusion
  * Stem cell mobilization will be performed for all subjects at the end of Cycle 4.
  Subjects may elect to stop E-RVD at the end of Cycle 4 and proceed to autologous SCT. Subjects who do not proceed to SCT may receive 8 cycles of induction therapy.
  The maintenance schedule (28 days) will start after 8 cycles of induction regimen for subjects not proceeding with SCT, or after recovery from SCT for subjects proceeding with it.
  Maintenance therapy with E-RVD will be administered to all patients, with the specific maintenance regimen determined by risk category.
Arm/Group | All Patients Treated With E-RVD.
Number analyzed (Participants) | 40
proportion of participants | 0.950 [0.831 to 0.994]

7. Secondary Outcome: Median Time to Response
Description: Time to response is defined as the time from the first dose of study drug to the first documentation of response partial response (PR) or better. Disease response was assessed using International Myeloma Working Group (IMWG) response criteria: Partial Response (PR) defined as 50% reduction of serum M-protein and reduction in 24h urinary M-protein by ≥90% or to <200mg/24h; Very Good Partial Response (VGPR) defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein plus urine M-protein level <100mg/24h; Complete Response (CR) defined as negative immunofixation on serum and urine and, disappearance of any soft tissue plasmacytomas and, <5% plasma cells in BM; Stringent Complete Response (sCR) defined as normal FLC ratio and absence of clonal cells in BM by immunohistochemistry or 2-4 color flow cytometry.
Time Frame: Participants were followed up to 92 days.
Population: This analysis population was restricted to the subjects whose best response was PR or better.
Measure: Median (Full Range); unit: days
Arm/Group | Elotuzumab, Lenalidomide, Bortezomib, and Dexamethasone
Number analyzed (Participants) | 38
days | 22.0 [20 to 92]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed every cycle on treatment, through study completion, an average of 6 years.
Arm/Group | Elotuzumab, Lenalidomide, Bortezomib, and Dexamethasone
All-Cause Mortality (participants affected / at risk) | 1/40
Serious Adverse Events (participants affected / at risk) | 10/40
Other Adverse Events (participants affected / at risk) | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elotuzumab, Lenalidomide, Bortezomib, and Dexamethasone (N=40)
Cardiac arrest (Cardiac disorders) | 1
Demyelating polyneuropathy (Nervous system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hyperglycemia (Endocrine disorders) | 1
Hypocalcemia (General disorders) | 1
Mood change (Psychiatric disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Pain in back (Musculoskeletal and connective tissue disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Blood and lymphatic system disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elotuzumab, Lenalidomide, Bortezomib, and Dexamethasone (N=40)
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Anemia (Blood and lymphatic system disorders) | 4
Fatigue (General disorders) | 23
Constipation (Gastrointestinal disorders) | 18
Peripheral neuropathy (Nervous system disorders) | 18
Diarrhea (Gastrointestinal disorders) | 12
Insomnia (Psychiatric disorders) | 12
Pain in back (Musculoskeletal and connective tissue disorders) | 12
Hypophosphatemia (Investigations) | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 9
Hyperglycemia (Investigations) | 9
Nausea (Gastrointestinal disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 8
Edema limbs (General disorders) | 7
Edema peripheral (General disorders) | 7
Transaminitis (Investigations) | 7
Blurred vision (Eye disorders) | 6
Headache (Nervous system disorders) | 6
Cramping in extremities (Musculoskeletal and connective tissue disorders) | 5
Fever (General disorders) | 5
Hypertension (General disorders) | 5
Mood change (Psychiatric disorders) | 5
Anxiety (Psychiatric disorders) | 4
Dry mouth (Gastrointestinal disorders) | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Hypotension (General disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in neck (Musculoskeletal and connective tissue disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Congestion (General disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Erythema at injection site (Skin and subcutaneous tissue disorders) | 3
Hypokalemia (General disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 3
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Night sweats (General disorders) | 3
Orthostatic hypotension (General disorders) | 3
Pruritis (Skin and subcutaneous tissue disorders) | 3
Stomach pain (Gastrointestinal disorders) | 3
Syncope (Nervous system disorders) | 3
Thrush (Infections and infestations) | 3
Tremor (Nervous system disorders) | 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3
Bruising (Skin and subcutaneous tissue disorders) | 2
Cataract (Eye disorders) | 2
Chest pain (Cardiac disorders) | 2
Chills (General disorders) | 2
Confusional state (Nervous system disorders) | 2
Decreased appetite (General disorders) | 2
Decreased magnesium (General disorders) | 2
Deep vein thrombosis (Cardiac disorders) | 2
Dehydration (General disorders) | 2
Depression (Psychiatric disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Flushing (General disorders) | 2
Gait disturbance (General disorders) | 2
Hiccups (General disorders) | 2
Hot flush (General disorders) | 2
Hyperuricemia (General disorders) | 2
Hypocalcemia (General disorders) | 2
Hyponatremia (General disorders) | 2
Increased amylase (General disorders) | 2
Increased lipase (General disorders) | 2
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2
Macroglossia (General disorders) | 2
Muscle cramping (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Neuropathy (Nervous system disorders) | 2
Edema face (General disorders) | 2
Oropharyngeal pain (Gastrointestinal disorders) | 2
Pain in bone (Musculoskeletal and connective tissue disorders) | 2
Pain in feet (Musculoskeletal and connective tissue disorders) | 2
Pain in hips (Musculoskeletal and connective tissue disorders) | 2
Pain in legs (Musculoskeletal and connective tissue disorders) | 2
Pain in ribs (Musculoskeletal and connective tissue disorders) | 2
Pain in shoulders (Musculoskeletal and connective tissue disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 2
Sciatica (Nervous system disorders) | 2
Tachycardia (Cardiac disorders) | 2

LIMITATIONS AND CAVEATS:
Limitations include lack of comparator arm. Small sample size; unable to draw valid conclusions from comparison studies. Duration of follow-up was limited and longer-term assessment of patient safety is warranted. Tolerability data is limited as patient-reported outcomes data not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT02375555/Prot_SAP_000.pdf